CLINICAL TRIAL: NCT03228537
Title: A Feasibility Trial of Neoadjuvant Cisplatin-Pemetrexed With Atezolizumab in Combination and in Maintenance for Resectable Malignant Pleural Mesothelioma
Brief Title: Atezolizumab, Pemetrexed Disodium, Cisplatin, and Surgery With or Without Radiation Therapy in Treating Patients With Stage I-III Pleural Malignant Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01230; NCI-2017-01230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1619 (Other: SWOG); S1619 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-07-24; First posted 2017-07-25 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Biphasic Mesothelioma; Epithelioid Mesothelioma; Stage I Pleural Malignant Mesothelioma AJCC v7; Stage IA Pleural Malignant Mesothelioma AJCC v7; Stage IB Pleural Malignant Mesothelioma AJCC v7; Stage II Pleural Malignant Mesothelioma AJCC v7; Stage III Pleural Malignant Mesothelioma AJCC v7
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — atezolizumab; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Pemetrexed; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, surgery, RT) (Experimental): NEOADJUVANT: Patients receive atezolizumab IV over 30-60 minutes, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 2 hours on day 1. Cycles repeats every 21 days for 4 cycles in the absence of disease progression or unexpected toxicity.
  SURGERY: Within 21-90 days after completion of neoadjuvant therapy, patients undergo EPP or PD. Patients who undergo EPP will then undergo RT.
  MAINTENANCE: Within 90 days after completion of either PD or radiation (post-EPP), patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Procedure: Extrapleural Pneumonectomy; Drug: Pemetrexed Disodium; Procedure: Pleurectomy; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Extrapleural Pneumonectomy — Undergo EPP
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Procedure: Pleurectomy — Undergo PD
  Other Names: Excision of Pleura
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I pilot trial studies how well atezolizumab, pemetrexed disodium, cisplatin, and surgery with or without radiation therapy works in treating patients with stage I-III pleural malignant mesothelioma. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving atezolizumab, pemetrexed disodium, and cisplatin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving atezolizumab after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate if the regimen of neoadjuvant cisplatin-pemetrexed disodium (pemetrexed)-atezolizumab, surgery +/- radiation, then maintenance atezolizumab is feasible and safe for patients with resectable malignant pleural mesothelioma.

SECONDARY OBJECTIVES:

I. To evaluate progression free survival (both by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 and also using a modified RECIST for pleural tumors) in patients with resectable malignant pleural mesothelioma treated with a regimen of neoadjuvant cisplatin-pemetrexed-atezolizumab, surgery +/- radiation, followed by one year of maintenance atezolizumab.

II. To evaluate overall survival in patients with resectable malignant pleural mesothelioma treated with a regimen of neoadjuvant cisplatin-pemetrexed-atezolizumab, surgery +/- radiation, followed by one year of maintenance atezolizumab.

III. To evaluate response rate (confirmed and unconfirmed, complete and partial, both by RECIST 1.1 and also using a modified RECIST for pleural tumors) in the subset of this patient population with measurable disease.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate the association between immunohistochemical (IHC) expression of PD-L1 in tumors and clinical outcomes in mesothelioma patients treated with trimodality/bimodality therapy including atezolizumab (anti-PD-L1).

II. To evaluate the association between expression of immune-related genes identified by Immune Nanostring (depending on ribonucleic acid [RNA] availability) and clinical outcomes in mesothelioma patients treated with trimodality/bimodality therapy including atezolizumab.

III. To evaluate the association between multiplex immunofluorescence (IF) of up to 10 immune markers in two panels and clinical outcomes in mesothelioma patients treated with trimodality/bimodality therapy including atezolizumab.

OUTLINE:

NEOADJUVANT: Patients receive atezolizumab intravenously (IV) over 30-60 minutes, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 2 hours on day 1. Cycles repeats every 21 days for 4 cycles in the absence of disease progression or unexpected toxicity.

SURGERY: Within 21-90 days after completion of neoadjuvant therapy, patients undergo extrapleural pneumonectomy (EPP) or pleurectomy/decortication (PD). Patients who undergo EPP will then undergo radiation therapy (RT).

MAINTENANCE: Within 90 days after completion of either PD or radiation (post-EPP), patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: NEOADJUVANT
* Patient must have stage I-III malignant pleural mesothelioma that is deemed resectable and must be planning to undergo pleurectomy decortication (P/D) or extrapleural pneumonectomy (EPP)
* Patient must have epithelioid or biphasic histology (sarcomatoid histology is excluded); histologic diagnosis and typing of mesothelioma requires at least a core needle biopsy or surgical biopsy of the pleura via thoracoscopy and small thoracotomy; cytology only will not be regarded as sufficient for the diagnosis
* Patient must have computed tomography (CT) chest/abdomen/pelvis with contrast or fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/CT scan performed within 28 days prior to step 1 registration
* Patients must have non-measurable or measurable disease documented by CT or magnetic resonance imaging (MRI); the CT from a combined PET/CT may be used to document only non-measurable disease unless it is of diagnostic quality; measurable disease must be assessed within 28 days prior to step 1 registration; non-measurable disease must be assessed within 42 days prior to step 1 registration; all disease must be assessed and documented on the RECIST 1.1 and modified RECIST baseline tumor assessment form
* Patient must have undergone extended surgical staging including mediastinoscopy or endobronchial ultrasound; at minimum, samples must be obtained from the mediastinal stations 4R, 7 (subcarinal), and 4L; this surgical staging must be performed within 42 days prior to step 1 registration; patient must be T1-3 and N0-N2 (single station)
* Patient must undergo video-assisted thoracoscopic surgery and diagnostic laparoscopy within 28 days prior to step 1 registration to rule out peritoneal disease spread
* Patient must have consultation with a surgeon within 21 days prior to step 1 registration; the surgeon must confirm that the patient's disease is resectable by pleurectomy decortication (P/D) or extrapleural pneumonectomy (EPP) and that the patient is an appropriate candidate for the surgical procedures
* Patient must not have had prior immunotherapy or chemotherapy for malignant pleural mesothelioma
* Patient must have Zubrod performance status 0 or 1 documented within 28 days prior to step 1 registration
* Patients requiring hearing aids or reporting hearing loss must have audiogram performed within 28 days prior to step 1 registration
* Patient must have not had any major surgery or radiation within 28 days prior to step 1 registration; diagnostic thoracotomies and laparoscopies are not considered major surgeries
* Patients must not have any anticancer therapy or investigational agent within 28 days prior to step 1 registration
* Absolute neutrophil count (ANC) >= 1,500/mcl (documented within 28 days prior to step 1 registration)
* Hemoglobin >= 9 g/dl (documented within 28 days prior to step 1 registration)
* Platelets >= 100,000/mcl (documented within 28 days prior to step 1 registration)
* Creatinine =< 1.5 x upper limit of normal (ULN) (documented within 28 days prior to step 1 registration)
* Creatinine clearance >= 45 ml/min (documented within 28 days prior to step 1 registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 28 days prior to step 1 registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (within 28 days prior to step 1 registration)
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Patients must not be pregnant or nursing due to the potential teratogenic side effects of the protocol treatment; women of reproductive potential and men must have agreed to use an effective contraceptive method for the duration of study treatment and for 5 months (150 days) after the last dose of atezolizumab; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patient must NOT have a history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patient must NOT have a known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Patients must not have severe infections within 28 days prior to step 1 registration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Patients must not have active autoimmune disease that has required systemic treatment in past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; autoimmune diseases include, but are not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis; this protocol includes an immunotherapy agent which can precipitate known autoimmune diseases
* Patients must not have undergone prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patient must not have active tuberculosis
* Patient must not have history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis; this protocol includes an immunotherapy agent which can precipitate known pneumonitis
* Patient must not have active (chronic or acute) hepatitis B virus (HBV) infection as evidenced by testing performed within 28 days prior to registration; patients with past or resolved HBV infection are eligible; active HBV is defined as having a positive hepatitis B surface antigen (HBsAg) test; past or resolved HBV is defined as having a negative HBsAG test and a positive total hepatitis B core antibody (HBcAb) test; patient must not have active hepatitis C virus (HCV) infection as evidenced by testing performed within 28 days prior to registration; active HCV is defined as having a positive HCV antibody test followed by a positive HCV RNA test
* Patient must NOT have a known positive test for human immunodeficiency virus (HIV); patients do not need to be screened for HIV; patients with HIV are excluded due to a potential incompetent immune system and need for medications that could interfere with the treatment and immunotherapy
* Patient must not have significant cardiovascular disease, such as New York Heart Association cardiac disease (class II or greater), myocardial infarction within 3 months prior to initiation of treatment, unstable arrhythmias, or unstable angina given the higher risks associated with surgical resection
* Patient must not receive live, attenuated influenza vaccine within 4 weeks prior to registration or at any time during the study and until 5 months after the last dose of atezolizumab
* Patient must be willing to have tissue specimens submitted for translational medicine studies
* Patient must be offered the opportunity to participate in tissue and blood banking for future studies
* Patient must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2: SURGERY
* Patient must have a CT of chest/abdomen with contrast or FDG-PET/CT scan within 28 days prior to step 2 registration; patients must not have evidence of progression per RECIST 1.1 or modified RECIST for pleural tumors
* Patients planning to receive EPP must also be evaluated for appropriateness of radiation therapy (RT) by a radiation oncologist within 14 days prior to step 2 registration
* Patients must have a Zubrod performance status of 0-1 documented within 28 days prior to step 2 registration
* Patients must have postoperative predicted forced expiratory volume in 1 second (FEV1) > 35% prior to surgery obtained within 28 days prior to step 2 registration; pulmonary function tests to ascertain these values must be obtained within 28 days prior to Step 2 registration
* Patients must have postoperative predicted carbon monoxide diffusing capability (DLCO) > 35% prior to surgery obtained within 28 days prior to step 2 registration; pulmonary function tests to ascertain these values must be obtained within 28 days prior to Step 2 registration
* Patient must have received at least two cycles of triplet neoadjuvant therapy (all three drugs) during step 1
* Patient must be registered to step 2 no less than 21 days and no more than 90 days after the end of their final cycle of neoadjuvant therapy
* STEP 3: MAINTENANCE
* Patient must have received either P/D or EPP and must have recovered from all effects of surgery with adequate wound healing; patients who received radiation therapy (RT) must be registered to step 3 within 90 days after discontinuing RT; patients who did not receive RT must be registered to step 3 within 90 days after surgery
* Patient must have a CT of chest/abdomen/pelvis with contrast or FDG-PET/CT scan within 28 days prior to step 3 registration; patient must not have evidence of progression per RECIST 1.1 or modified RECIST for pleural tumors
* Patient may have discontinued RT early due to toxicity or other reasons
* Patients must have a Zubrod performance status of 0-1 documented within 28 days prior to step 3 registration
* ANC > 1,500/mcl (documented within 28 days prior to step 3 registration)
* Hemoglobin > 9 g/dl (documented within 28 days prior to step 3 registration)
* Platelets > 100,000/mcl (documented within 28 days prior to step 3 registration)
* Creatinine < 1.5 x ULN (documented within 28 days prior to step 3 registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 28 days prior to step 3 registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (within 28 days prior to step 3 registration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2026-09-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — SWOG Cancer Research Network
Locations (177):
- United States (177):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants were registered to the study, 1 participant was ineligible, so 28 participants received protocol treatment for Step 1, Neoadjuvant.
Groups:
- Treatment (Chemotherapy, Surgery +/- RT, Maintenance): NEOADJUVANT: Patients receive atezolizumab IV over 30-60 minutes, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 2 hours on day 1. Cycles repeats every 21 days for 4 cycles in the absence of disease progression or unexpected toxicity.
  SURGERY: Within 21-90 days after completion of neoadjuvant therapy, patients undergo extrapleural pneumonectomy (EPP) or pleurectomy/decortication (PD). Patients who undergo EPP will then undergo radiation therapy.
  MAINTENANCE: Within 90 days after completion of either PD or radiation (post-EPP), patients receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unexpected toxicity.
Period: Neoadjuvant
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Started | 28
Completed | 21
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Progression/Relapse | 4
Not completed — Death | 1
Period: Surgery
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Started | 19
Completed | 16
Not Completed | 3
Not completed — Death | 1
Not completed — Other - Not Protocol Specified | 2
Period: Maintenance
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Started | 15
Completed | 4
Not Completed | 11
Not completed — Refusal Unrelated to Adverse Event | 1
Not completed — Progression/Relapse | 10

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 68.1 [31.5 to 77.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic: No | 27
  Hispanic: Unknown | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 24
  Race: Asian | 3
  Race: Unknown | 1
Surgery [Count of Participants; unit: Participants]
  Extrapleural Pneumonectomy (EPP) | 4
  Pleurectomy/Decortication (PD) | 24
Performance Status [Count of Participants; unit: Participants] — Performance Status uses the Zubrod Scale as follows:
  0 - Fully active, able to carry on all pre-disease performance w/o restriction
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  Participants
    0 | 15
    1 | 13
Weight Loss Past 6 Months [Count of Participants; unit: Participants]
  <6% | 23
  5-<10% | 4
  Pending | 1
Baseline Disease Status mRECIST [Count of Participants; unit: Participants]
  Measurable | 22
  Not Assessable | 6
Baseline Disease Status RECIST [Count of Participants; unit: Participants]
  Measurable | 14
  Non-Measurable | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Neoadjuvant Cisplatin-Pemetrexed-Atezolizumab, Surgery +/- Radiation, and Maintenance Therapy.
Description: The number of participants who received at least two cycles of the triplet neoadjuvant therapy getting at least one dose of maintenance therapy.
Time Frame: Duration of treatment until first dose of maintenance therapy. Includes 21 day cycles of neoadjuvant chemo and surgery - extrapleural pneumonectomy or pleurectomy/decortication (radiation therapy for participants who received extrapleural pneumonectomy).
Population: Participants that received at least 2 cycles of neoadjuvant Cisplatin-Pemetrexed-Atezolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 25
Participants | 15

2. Primary Outcome: Safety of Neoadjuvant Cisplatin-Pemetrexed-Atezolizumab, Surgery +/- Radiation, and Maintenance Therapy.
Description: The number of participants that experienced a Grade 4-5 immune-related adverse event. The regimen was considered safe if no participants experienced a Grade 4-5 immune-related AE.
Time Frame: Duration of treatment and follow-up until death or 3 years post Step 1 registration.
Population: Participants who were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 28
Participants | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: From date of registration to Step 1 to date of first documentation of progression by RECIST 1.1 and modified RECIST 1.1, symptomatic deterioration, or death due to any cause. Participants last known to be alive and progression free are censored at date of last disease assessment.
Time Frame: Duration of treatment and follow-up until death or 3 years post Step 1 registration.
Population: Eligible and evaluable participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 28
Months
  RECIST 1.1 | 9.5 [6.6 to 13.0]
  mRECIST 1.1 | 18.4 [6.6 to 25.1]

4. Secondary Outcome: Overall Survival (OS)
Description: From date of initial registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: 3 years after the last accrual
Population: Eligible and evaluable participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 28
Months | 31.5 [18.4 to NA] — Less than half of the remaining participants died (more than half are still alive) after reaching the median survival.

5. Secondary Outcome: Response Rate (RR)
Description: Percentage of participants with confirmed and unconfirmed, complete and partial, defined by RECIST 1.1 and mRECIST for Pleural Tumors
Time Frame: Duration of treatment and follow-up until death or 3 years post Step 1 registration.
Population: Eligible and evaluable participants with measurable disease. 14 participants had measurable disease according to the RECIST which measures lesions from an x-ray, CT, or MRI. 22 participants had measurable disease according to the mRECIST which measures lesions as the sum of 6 CT cuts.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Surgery +/- RT, Maintenance)
Number analyzed (Participants) | 22
Participants
  RECIST 1.1: number analyzed (Participants) | 14
  RECIST 1.1 | 7
  mRECIST 1.1 | 10

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration to Step 1.
Description: CTCAE version 5.0 was used for reporting SAEs and routine toxicity reporting. There were 28 participants on registration Step 1 (Neoadjuvant) that were assessed for AEs, 19 participants on registration Step 2 (Surgery) that were assessed for AEs, and 15 participants on registration Step 3 (Maintenance) that were assessed for AEs.
Groups:
- Chemotherapy + Atezolizumab: Participants receive atezolizumab IV over 30-60 minutes, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 2 hours on day 1. Cycles repeats every 21 days for 4 cycles in the absence of disease progression or unexpected toxicity.
- Surgery: Within 21-90 days after completion of neoadjuvant therapy, participants undergo EPP or PD. Participants who undergo EPP will then undergo RT.
- Maintenance: Within 90 days after completion of either PD or radiation (post-EPP), participants receive atezolizumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 1 year in the absence of disease progression or unexpected toxicity.
Arm/Group | Chemotherapy + Atezolizumab | Surgery | Maintenance
All-Cause Mortality (participants affected / at risk) | 6/28 | 3/19 | 6/15
Serious Adverse Events (participants affected / at risk) | 11/28 | 0/19 | 2/15
Other Adverse Events (participants affected / at risk) | 28/28 | 16/19 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Atezolizumab (N=28) | Surgery (N=19) | Maintenance (N=15)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0
Infusion related reaction (General disorders) | 3 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Atezolizumab (N=28) | Surgery (N=19) | Maintenance (N=15)
Anemia (Blood and lymphatic system disorders) | 13 | 9 | 10
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0 | 2
Blurred vision (Eye disorders) | 1 | 1 | 1
Eye disorders-Other (Eye disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 11 | 2 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 21 | 3 | 7
Vomiting (Gastrointestinal disorders) | 7 | 3 | 2
Chills (General disorders) | 1 | 0 | 1
Edema limbs (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 16 | 5 | 11
Fever (General disorders) | 4 | 0 | 2
General disorders and admin site conditions - Other (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 4 | 6
Pain (General disorders) | 2 | 5 | 4
Lung infection (Infections and infestations) | 1 | 0 | 2
Pleural infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Creatinine increased (Investigations) | 6 | 5 | 4
Lymphocyte count decreased (Investigations) | 5 | 0 | 2
Neutrophil count decreased (Investigations) | 11 | 0 | 0
Platelet count decreased (Investigations) | 2 | 3 | 2
Weight gain (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 2 | 2 | 0
White blood cell decreased (Investigations) | 8 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 12 | 4 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 3 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 5 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 1 | 2
Dysgeusia (Nervous system disorders) | 6 | 1 | 0
Headache (Nervous system disorders) | 8 | 1 | 2
Paresthesia (Nervous system disorders) | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 4 | 0 | 2
Hypotension (Vascular disorders) | 2 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03228537/Prot_SAP_000.pdf